CLINICAL TRIAL: NCT05389163
Title: Clinical Evaluation of Giomer Based Injectable Resin Composite Versus Resin Modified Glass Ionomer in Class V Carious Cavities Over 18-months: Randomized Controlled Trial
Brief Title: Clinical Evaluation of Giomer Based Injectable Resin Composite Versus Resin Modified Glass Ionomer in Class V Carious Cavities Over 18-months.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Adel Yahia Hendam, assistant lecturer at conservative department,,faculty of dentistry, modern university for Technology and Information., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Giomer vs RMGI in class V
Record Dates: First submitted 2022-05-12; First posted 2022-05-25 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Class V Dental Caries
Keywords: Giomer; injectable resin composite; Resin modified glass ionomer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Giomer based injectable resin composite (Experimental): Beautifil Flow plus X F03, SHOFU, USA
  Interventions: Device: Giomer based injectable resin composite
- Resin modified glass ionomer (Active Comparator): Fuji II LC, GC
  Interventions: Device: Resin modified glass ionomer

INTERVENTIONS:
Device: Giomer based injectable resin composite — Giomer material has been introduced as the true hybridization of glass ionomer and resin composite, containing surface pre-reacted glass ionomer (S-PRG) filler particles within a resin matrix. Giomer combines caries protection through fluoride release and recharge of glass ionomers and the esthetics, physical and handling properties of resin composite
  Arms: Giomer based injectable resin composite
Device: Resin modified glass ionomer — Resin modified glass ionomer (RMGI) have been developed to combine the advantages of both resin composite and glass ionomer; the good mechanical properties, esthetic of resin composite added to anticariogenic activity and chemical bonding to tooth structure of glass Ionomer.
  Arms: Resin modified glass ionomer

SUMMARY:
Class V carious lesions will be restored using either Resin modified glass ionomer or Giomer based injectable resin composite.The restorations will be evaluated at baseline and regular recalls of 3 months, 6 months, 12 months and 18 months, using modified United States Public Health Service criteria.

DETAILED DESCRIPTION:
In this study, Class V carious lesions will be restored using two different restorative materials either Resin modified glass ionomer or Giomer based injectable resin composite. Patients will be assessed for medical and dental histories first. Then an examination of the patients will be done using visual inspection by using a dental mirror and probe. Eligible patients according to inclusion and exclusion criteria will be informed about all procedures with follow up time if they accept. Their signature on written informed consents will be obtained. Eligible participants will be randomly divided into two groups according to the type of restoration they will be received.The first group (A) (Intervention): Giomer based injectable resin composite (Beautifil Flow plus X F03, SHOFU, USA): The material will be applied according to manufacturer instructions. The second group (B) (comparator): Resin modified glass ionomer (Fuji II LC, GC): The material will be applied according to manufacturer instructions.The restorations will be evaluated at baseline and regular recalls of 3 months, 6 months, 12 months and 18 months, using modified United States Public Health Service criteria (USPHS) for the following characteristics: retention, anatomical form, marginal adaptation, marginal staining, surface texture, and secondary caries . The restorations will be evaluated with the aid of a dental explorer and an intraoral mirror and visual inspection. The restorations will be scored as follows: Alfa represents the ideal clinical situation, Bravo will be clinically acceptable, and Charlie represents a clinically unacceptable situation.

ELIGIBILITY:
Participant Inclusion Criteria

* Age 18-60 years.
* Co-operative patients approving to participate in the study.
* Male or female patients.
* Patients with good general health
* Moderate or high caries risk patient

Teeth Inclusion Criteria

* Cervical Class V carious lesions.
* Pulp asymptomatic vital carious teeth.

Participant Exclusion Criteria

* Systemic disease or severe medical complications.
* Participants with a history of allergy to any component of restorations will be used in the study.
* Lack of compliance
* Evidence of severe bruxism, clenching, or temporomandibular joint disorders or bizarre habits

Teeth Exclusion Criteria

* Presence of apical or periapical pathosis.
* tooth mobility
* Non-vital teeth.
* Teeth with advanced periodontal diseases.
* Teeth which need indirect restoration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Clinical performance (Marginal adaptation) | 18 months
  Method of measurement is Modified United State Public Health Service Criteria (Modified USPHS) using (Alpha, Bravo, charlie) as unit of measurement by Scoring %.
  Alpha is the best outcome and charlie is the worse outcome .

SECONDARY OUTCOMES:
Clinical performance (Anatomical form, marginal discoloration, Secondary caries, surface texture , Postoperative sensitivity, Retention,) | 18 months
  Method of measurement is Modified United State Public Health Service Criteria (Modified USPHS) using (Alpha, Bravo, charlie) as unit of measurement by Scoring %.
  Alpha is the best outcome and charlie worse outcome .

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Expecting to have all the data by October 2024